CLINICAL TRIAL: NCT01444352
Title: Study of an Investigational Pneumococcal Vaccine at Three Dose Levels in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PPR06
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Pneumococcal Infections; Streptococcus Pneumoniae Infections; Pneumococcal Pneumonia
Keywords: Pneumococcal infections; Streptococcus pneumoniae Infections; Pneumococcal Vaccines
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia, Pneumococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vaccine Formulation 1 (Low dose) (Experimental): Participants will receive 2 injections of Pneumococcal Vaccine Formulation 1 (Low dose).
  Interventions: Biological: Pneumococcal vaccine Formulation 1
- Vaccine Formulation 2 (Middle dose) (Experimental): Participants will receive 2 injections of Pneumococcal Vaccine Formulation 2, (Middle dose).
  Interventions: Biological: Pneumococcal vaccine Formulation 2
- Vaccine Formulation 3 (High dose) (Experimental): Participants will receive 2 injections of Pneumococcal Vaccine Formulation 3, (High dose).
  Interventions: Biological: Pneumococcal vaccine Formulation 3
- Placebo Pooled (Placebo Comparator): Participants who receive 2 injections of tris buffered saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Pneumococcal vaccine Formulation 1 — 0.5 mL, Intramuscular (Low dose)
  Arms: Vaccine Formulation 1 (Low dose)
Biological: Pneumococcal vaccine Formulation 2 — 0.5 mL, Intramuscular (Middle dose)
  Arms: Vaccine Formulation 2 (Middle dose)
Biological: Pneumococcal vaccine Formulation 3 — 0.5 mL, Intramuscular (High dose)
  Arms: Vaccine Formulation 3 (High dose)
Biological: Placebo — 0.5 mL, Intramuscular
  Other Names: Tris Buffered Saline
  Arms: Placebo Pooled

SUMMARY:
This study is designed to evaluate the safety, tolerability, and immunogenicity of an investigational pneumococcal vaccine in healthy adult volunteers.

Primary Objective:

* To evaluate the safety and tolerability of an investigational pneumococcal vaccine.

Observational Objective:

* To evaluate the immunogenicity of an investigational Pneumococcal vaccine.

DETAILED DESCRIPTION:
An initial cohort of 10 participants will receive a single dose of investigational pneumococcal vaccine. After safety assessment of this cohort during a 24-hour in-unit observation period, additional cohorts will receive two injections of the study vaccine 30 days apart, at three dose levels, in ascending doses by cohort, pending safety review at each dose level. All participants will be monitored for safety for 30 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and comply with all trial procedures
* Subject is healthy, as determined by medical history and physical examination
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to first vaccination until 4 weeks after the last vaccination.

Exclusion Criteria:

* History of anaphylactic reaction or asthma
* Unknown pregnancy or positive serum/urine pregnancy test
* Currently breastfeeding a child
* Chronic illness, that in the opinion of the investigator, is at a stage that could interfere with trial conduct or completion
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, except for pandemic influenza vaccination which may be received at least two weeks before the study vaccines
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination, except for pandemic influenza vaccination in the event of a local or national immunization program
* Known seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Laboratory confirmed/self-reported thrombocytopenia contraindicating intramuscular (IM) vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as a study site employee who is involved in the protocol and may have direct access to trial-related data
* Previous vaccination against pneumococcal disease (in the previous 5 years)
* History of pneumococcal infection (confirmed either clinically, serologically, or microbiologically) within 5 years
* At high risk for pneumococcal infection during the trial
* Living in a household with children <5 years of age.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants reporting solicited injection site reactions, solicited systemic reactions, unsolicited systemic reactions, and serious adverse events occurring throughout the trial | Days 0 through 30 post-vaccination
  Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.

SECONDARY OUTCOMES:
Immunogenicity of Pneumococcal Vaccine After two Vaccinations | Days 0 and 30 days post-vaccination
  Evaluation of immune responses to antigen component of the investigational vaccine by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Ltd.
Locations (1):
- Allschwil, Switzerland

REFERENCES:
- [Derived] Kamtchoua T, Bologa M, Hopfer R, Neveu D, Hu B, Sheng X, Corde N, Pouzet C, Zimmermann G, Gurunathan S. Safety and immunogenicity of the pneumococcal pneumolysin derivative PlyD1 in a single-antigen protein vaccine candidate in adults. Vaccine. 2013 Jan 2;31(2):327-33. doi: 10.1016/j.vaccine.2012.11.005. Epub 2012 Nov 12. PMID 23153437
- See also: Related Info — http://www.sanofipasteur.com